CLINICAL TRIAL: NCT03200054
Title: Postpartum Adherence Clubs for Antiretroviral Therapy: a Randomised Controlled Trial
Brief Title: Postpartum Adherence Clubs for Antiretroviral Therapy
Acronym: PACART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Professor Landon Myer, Head: Department of Public Health and Family Medicine, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 195/2015
Record Dates: First submitted 2017-03-21; First posted 2017-06-27 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Hiv
Keywords: therapy; postnatal
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinic-based Care (No Intervention): Clinic-based care is the current standard of care and is defined as referral of women on antiretroviral therapy (ART) to general primary care adult ART services.
- Adherence Club Care (Experimental): Adherence club care involves referral of women on ART to community-based ART services in the form of adherence clubs, which are led by community health workers and supported by ART clinic nurses.
  Interventions: Other: Adherence Clubs

INTERVENTIONS:
Other: Adherence Clubs — Women will be referred to the ACs at their postpartum ART clinic visit at the midwife obstetric unit (MOU) at the Gugulethu community health centre (CHC). AC visits occur 2-4 monthly at a community hall near the CHC. At routine visits, which last ~1 hour, community health workers provide health education, weigh participants, ask about symptoms, and dispense pre-packed ART. Symptomatic participants are referred back to the main ART facility at the CHC for assessment by a nurse. A nurse performs routine phlebotomy at an annual club visit, and does a clinical assessment and reviews blood results at the subsequent visit. Participants requiring more regular follow-up and those with raised viral loads are referred back to the ART clinic at the CHC by the nurse.
  Arms: Adherence Club Care

SUMMARY:
South Africa is implementing the policy of universal initiation of lifelong antiretroviral therapy (ART) in all HIV-infected pregnant women regardless of CD4 cell count or disease stage ("Option B+"). There is a recognised need for innovative models of service delivery to support adherence and retention in care in this group, particularly during the postpartum period. The investigators are conducting a pragmatic randomised control trial to compare virological outcomes 24 months postpartum in two models of service delivery for provision of HIV care and treatment services postpartum in women who initiated ART during pregnancy: local adult ART clinics and community-based adherence clubs.

DETAILED DESCRIPTION:
South Africa is implementing the policy of universal initiation of lifelong ART in all HIV-infected pregnant women regardless of CD4 cell count or disease stage ("Option B+") and given the high antenatal HIV seroprevalence, HIV-infected pregnant women represent the largest group of patients initiating ART in primary care facilities. However, there are few well developed models of service delivery to support implementation. There are particular concerns regarding the postpartum period, with multiple studies indicating high levels of non-retention in care and/or inadequate adherence to treatment postnatally. Adherence Clubs (ACs) are an innovative but untested model of care based on chronic disease management strategies that emphasize social support, adherence to treatment and retention in care, rather than intensive clinical management, as the most important determinant of long-term health outcomes in stable patients in chronic care. ACs have preliminarily been shown to to result in virologic outcomes that are similar to routine clinic services in patients stable on ART. The investigators are conducting a pragmatic, randomised controlled trial to evaluate two different strategies for delivering HIV care and treatment services during the postpartum period to HIV-infected women who initiated ART during pregnancy. Participants will be allocated to receive ART care at either local adult ART clinics, following the current standard of care, or the community-based adherence club system.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection with ART initiation during the preceding antenatal period
* Within 70 days post-delivery
* Viral suppression documented in pregnancy with the most recent viral load <400 copies/mL within the last 3 months
* Willingness to be randomised and return for study measurement visits
* Able and willing to attend service visits at either a local ART treatment centre or the adherence club at Ikhwezi centre
* Able to provide informed consent for research

Exclusion Criteria:

* Intention to relocate out of Cape Town permanently during the study period
* Any medical, psychiatric or social condition which in the opinion of the investigators would affect the ability to consent and/or participate in the study including: refusal to take ART/antiretrovirals (ARVs) and/or denial of HIV status
* Loss of pregnancy/neonate at the time of eligibility determination
* Current co-morbidity requiring additional health care attention, including opportunistic infections such as tuberculosis (TB) disease or any chronic condition or other condition that is not controlled or stable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Viral suppression | 24 months
  Time to viral load >1000 copies per ml

SECONDARY OUTCOMES:
Maternal retention in care | 24 months
  Missed routinely scheduled clinical care visits (missed visit and no visit within 3 months of scheduled clinic visit)
Maternal death | 24 months
  Maternal deaths over the study period
Maternal mental health | 24 months
  Mental health as assessed via brief screening tools (Edinburgh Postnatal Depression Scale)
Maternal health care service use | 24 months
  Use of health facilities including hospitalization
Infant death | 24 months
  Infant deaths over the study period
Infant health care service use | 24 months
  Use of health facilities including hospitalization
Infant HIV testing | 24 months
  Uptake of routine infant HIV testing
Infant HIV infection | 24 months
  Mother-to-child transmission of HIV
Infant feeding | 24 months
  Breastfeeding practices
Cost and cost-effectiveness | 24 months
  Cost-effectiveness of each strategy will be analysed from both the patient and health systems perspective
Acceptability of each ART service | 24 months
  Acceptability of each service will be assessed using the patient-provider interview schedule, and qualitative interviews will be done on a subset of participants
Viral suppression at other cutpoints (>400 copies/mL) | 24 months
  Time to VL >400 copies/mL
Viral suppression at other cutpoints (>50 copies/mL) | 24 months
  Time to VL >50 copies/mL
Virologic Failure | 24 months
  Time to clinical definition of virologic failure (two consecutive VLs >1000 copies/mL)
Combined retention/VL outcome | 24 months
  Composite endpoint of retention in care and viral suppression (not retained in care OR retained but VL >50 or 1000 copies/mL)
Viral suppression at each study visit | 24 months
  VL >50 copies/mL or >1000 copies/mL at each study visit (3, 6, 12, 18, 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Landon Myer, MBChB PhD, Principal Investigator — University of Cape Town
Locations (1):
- Gugulethu Community Health Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan R, Orrell C, Zwane E, Bekker LG, Wood R. Loss to follow-up and mortality among pregnant women referred to a community clinic for antiretroviral treatment. AIDS. 2008 Aug 20;22(13):1679-81. doi: 10.1097/QAD.0b013e32830ebcee. PMID 18670232
- [Background] Nachega JB, Uthman OA, Anderson J, Peltzer K, Wampold S, Cotton MF, Mills EJ, Ho YS, Stringer JS, McIntyre JA, Mofenson LM. Adherence to antiretroviral therapy during and after pregnancy in low-income, middle-income, and high-income countries: a systematic review and meta-analysis. AIDS. 2012 Oct 23;26(16):2039-52. doi: 10.1097/QAD.0b013e328359590f. PMID 22951634
- [Background] Coutsoudis A, Goga A, Desmond C, Barron P, Black V, Coovadia H. Is Option B+ the best choice? Lancet. 2013 Jan 26;381(9863):269-71. doi: 10.1016/S0140-6736(12)61807-8. No abstract available. PMID 23351797
- [Background] Chi BH, Stringer JS, Moodley D. Antiretroviral drug regimens to prevent mother-to-child transmission of HIV: a review of scientific, program, and policy advances for sub-Saharan Africa. Curr HIV/AIDS Rep. 2013 Jun;10(2):124-33. doi: 10.1007/s11904-013-0154-z. PMID 23440538
- [Background] Luque-Fernandez MA, Van Cutsem G, Goemaere E, Hilderbrand K, Schomaker M, Mantangana N, Mathee S, Dubula V, Ford N, Hernan MA, Boulle A. Effectiveness of patient adherence groups as a model of care for stable patients on antiretroviral therapy in Khayelitsha, Cape Town, South Africa. PLoS One. 2013;8(2):e56088. doi: 10.1371/journal.pone.0056088. Epub 2013 Feb 13. PMID 23418518
- [Background] Provincial Government of the Western Cape. PMTCT Clinical Guidelines Update, May 2013. Cape Town: PGWC; 2013.